CLINICAL TRIAL: NCT04825834
Title: DNA Evaluation of Fragments for Early Interception - Lung Cancer Training Study (DELFI-L101 Study)
Acronym: DELFI-L101
Status: Completed | Type: Observational
Sponsor: Delfi Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DELFI-L101 Study
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Head and Neck Cancer; Esophageal Cancer; Bladder Cancer; Kidney Cancer; Stomach Cancer; Colorectal Cancer; Pancreas Cancer; Liver Cancer; Skin Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood specimens may be used to develop and evaluate performance of biomarker assays to detect cancers or other conditions, laboratory process improvements, and proficiency testing. Residual blood specimens will be de-identified and will be stored for no more than 20 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Individuals eligible for Lung Cancer screening with Lung Cancer diagnosis
  Interventions: Other: Blood Sample Collection
- Individuals eligible for Lung Cancer screening with no cancer diagnosis
  Interventions: Other: Blood Sample Collection
- Individuals eligible for Lung Cancer screening with Non-Lung Cancer diagnosis
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects enrolled in the DELFI-L101 will have blood specimens collected (~40 mL) at enrollment.

SUMMARY:
The primary objective of this study, DELFI-L101, is to train and test classifiers for lung cancer detection using the DELFI assay and other biomarker and clinical features.

DETAILED DESCRIPTION:
Subjects will be enrolled into the DELFI-L101 study after informed consent and eligibility is confirmed. At enrollment, subjects will have blood specimens collected (~40 mL) and 12 months post-enrollment their medical records will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

1. Ability to understand and provide written informed consent
2. Age ≥ 50 years
3. Current or Former Smoker
4. ≥ 20 pack-years (pack years = number of packs per day X number of years smoked)

   Inclusion Group 1: High Risk Patients that meet criteria 5 and 6 below:
5. Prior thoracic imaging with computed tomography (CT) within 12 months of enrollment (CT imaging for lung cancer screening for participants meeting inclusion criteria 6a and 6b; or CT imaging for lung cancer screening or diagnostic CT for participants meeting inclusion criteria 6c)

   OR Planned thoracic imaging (CT) as part of standard of care within 6 weeks of enrollment (CT imaging for lung cancer screening for participants meeting inclusion criteria 6a and 6b; or CT imaging for lung cancer screening or diagnostic CT for participants meeting inclusion criteria 6c)

   AND
6. Meet one of the criteria below:

   1. No suspected or confirmed lung cancer diagnosis OR
   2. Suspected of lung cancer OR
   3. Confirmed, untreated lung cancer

   Inclusion Group 2: High Risk Patients that meet the following criteria:
7. Pathologic confirmed, invasive non-lung cancer diagnosis, originating from the esophagus (upper), colon or rectum, pancreas, stomach (including lower esophagus), head and neck, skin (excluding cutaneous basal cell and squamous cell carcinoma) kidney, or liver, with no prior systemic therapy, definitive therapy, radiation, or surgical resection.

OR Clinically confirmed invasive non-lung cancer diagnosis originating from the pancreas, kidney, or liver, based on imaging and clinical judgment with planned treatment and no prior systemic therapy, definitive therapy, radiation, or surgical resection.

OR Clinically (based on imaging and clinical judgment) or pathologically confirmed non-invasive or invasive bladder cancer with planned treatment and no prior systemic therapy, definitive therapy, radiation or surgical resection.

Exclusion Criteria:

All Participants:

1. Prior systemic therapy, definitive therapy, radiation, or surgical resection for cancer within one year prior to enrollment (with the exception of organ biopsies or surgery for non-melanoma skin cancer)
2. Any history of hematologic malignancies or myelodysplasia
3. Any history of organ tissue transplantation
4. Any history of blood product transfusion
5. Current pregnancy
6. Any condition that in the opinion of the Investigator should preclude the participant's participation in the study
7. Prior systemic therapy, definitive therapy, radiation, or surgical resection for the enrollment cancer diagnosis (with the exception of organ biopsies or surgery for non-melanoma skin cancer are not exclusionary)
8. Enrollment in any DELFI sponsored study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals ≥ 50 years of age who are eligible for lung cancer screening from medical, surgical, sub- specialty clinics, lung cancer screening, lung nodule, thoracic surgery, and chest clinic practices.
Sampling Method: Non-Probability Sample
Enrollment: 2992 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of lung cancer detection measured by sensitivity, specificity, and the AUC of the ROC. | Approximately 12 months

SECONDARY OUTCOMES:
Accuracy (sensitivity and specificity) in clinical subgroups of interest | Approximately 12 months
Prevalence-based measures, including positive predictive value (PPV), negative predictive value (NPV), and number needed to screen (NNS) | Approximately 12 months
Accuracy of tumor of origin (confusion matrix of predicted versus actual cancer type) | Approximately 12 months
Adverse events (AEs) associated with the blood specimen collection | Point in time of blood specimen collection (1day) at enrollment
Expected distribution of the DELFI score in the intended use population and clinical subgroups of interest | Approximately 12 months
Association of genomic features with clinical subgroups of interest | Approximately 12 months
Analytical performance (e.g. repeatability/reproducibility) | Approximately 12 months
Accuracy of multi-cancer detection measured by sensitivity, specificity, and the AUC of the ROC and tissue of origin (TOO) accuracy | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mazzone, MD, MPH, Principal Investigator — The Cleveland Clinic; Luke RG Pike, MD, DPhil, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (57):
- United States (56):
  - Central Alabama Research, Homewood, Alabama
  - Phoenix Medical Group, Peoria, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Pulmonary Associates of Burlingame, Burlingame, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Centura Health, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - St. Mary's Hospital and Regional Medical, Grand Junction, Colorado
  - Starling Physicians, New Britain, Connecticut
  - Stamford Health, Stamford, Connecticut
  - Baycare, Clearwater, Florida
  - Oncology & Hematology Associates of West Broward, Coral Springs, Florida
  - Holy Cross Hospital Cancer Center, Fort Lauderdale, Florida
  - Miami Cancer Institute, Miami, Florida
  - Charter Research - The Villages, Orlando, Florida
  - Millennium Physicians Group, LLC, Port Charlotte, Florida
  - Charter Research - The Villages, The Villages, Florida
  - Pulmonary and Sleep Specialists of Northeast Georgia - Dacula, Dacula, Georgia
  - Christie Clinic, Champaign, Illinois
  - Duly Health and Care, Joliet, Illinois
  - Edward-Elmhurst Healthcare, Naperville, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Louisville Pulmonary Care, PLLC, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Gulfport, Gulfport, Mississippi
  - Washington University at St. Louis, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Holy Name Pulmonary Associates, Englewood, New Jersey
  - Atlantic Digestive Health Institute, Morristown, New Jersey
  - Oncology Hematology Specialists, Mountain Lakes, New Jersey
  - MedCorps Asthma and Pulmonary Specialists - Sewell, Sewell, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Northwell Health, New York, New York
  - CHEAR Center LLC, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Respiratory Specialists, Ltd., Wyomissing, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Austin Regional Clinic ARC Clinical Research at Wilson Parke, Austin, Texas
  - Premier Family Physicians, Austin, Texas
  - Pulmonary Critical Care & Sleep Associates, P.A., Conroe, Texas
  - Huntsville Research Institute, LLC, Huntsville, Texas
  - ProHealth Care, Waukesha, Wisconsin
- Pan American Center for Oncology Trials, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzone PJ, Bach PB, Carey J, Schonewolf CA, Bognar K, Ahluwalia MS, Cruz-Correa M, Gierada D, Kotagiri S, Lloyd K, Maldonado F, Ortendahl JD, Sequist LV, Silvestri GA, Tanner N, Thompson JC, Vachani A, Wong KK, Zaidi AH, Catallini J, Gershman A, Lumbard K, Millberg LK, Nawrocki J, Portwood C, Rangnekar A, Sheridan CC, Trivedi N, Wu T, Zong Y, Cotton L, Ryan A, Cisar C, Leal A, Dracopoli N, Scharpf RB, Velculescu VE, Pike LRG. Clinical Validation of a Cell-Free DNA Fragmentome Assay for Augmentation of Lung Cancer Early Detection. Cancer Discov. 2024 Nov 1;14(11):2224-2242. doi: 10.1158/2159-8290.CD-24-0519. PMID 38829053